CLINICAL TRIAL: NCT04951271
Title: The Effect of Solution Focused Approach on Anger Management and Violent Behavior in Adolescents: A Randomized Controlled Trial
Brief Title: Anger Management and Violent Behavior in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, EBRU AKBAŞ, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Adolescent, anger management
Record Dates: First submitted 2021-06-23; First posted 2021-07-06 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Adolescent; Anger; Violent Behavior
Keywords: Solution Focused Approach; Adolescent; Anger Management; Violent Behavior; Psychiatric nursing

STUDY DESIGN:
Intervention Model Description: This research is a single-blind, randomized controlled study with a control group design with pre-test and post-test measurements from experimental research designs.
Who Masked: Participant, Outcomes Assessor
Masking Description: Which students were included in the experimental and control groups was determined by simple randomization. Thus, a one-way blinding was made by preventing the adolescent students included in the study from knowing whether they were in the experimental group or the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (SFA) group (Experimental): solution-focused approach intervention was applied for 7 weeks
  Interventions: Behavioral: Solution focused approach
- Control (no intervention) group (No Intervention): No intervention was made.

INTERVENTIONS:
Behavioral: Solution focused approach — The SFA intervention consists of seven sessions, one preparation and six solution-oriented sessions. Each session lasted 55 minutes. Filling in the applied scales was excluded from this period. Sessions were held once a week in two groups (Grade 10 and Grade 11 students).
  Arms: Intervention (SFA) group

SUMMARY:
The research was conducted to examine the effect of solution focused approach on anger management and violent behavior in adolescents.

DETAILED DESCRIPTION:
Anger, which is one of the universal emotions; It is a natural response to unsatisfied demands, frustrations, and unmet expectations. Adolescents are the group that most experience the feeling of anger that everyone frequently encounters in daily life.

Adolescent individuals may have more difficulty in controlling their anger than other age groups. Inappropriately expressed anger; It can lead to various physical, social and psychological problems such as incompatibility in interpersonal relationships, negative effects on health, disagreement in the workplace, conflict and violence.

Adolescents who do not know how to deal with their anger can engage in various violent behaviors by expressing their anger in inappropriate ways. Aggressive behaviors that develop due to the tendency of violence in young people pose a problem in terms of public health, considering the effects on the mental health and well-being of adolescents. In studies examining the victims of violence in the adolescent period; It has been determined that the victims have a wide range of health and psychological problems.

There are various approaches that support anger control psychosocially for adolescents, who are a risky group in anger control. Preventive intervention programs are implemented for adolescents on the causes of anger, anger expression patterns, anger management, problem solving techniques, improving communication skills and stress management. Recently, Solution-Focused Approach (SFA), which is one of the alternative approaches that focuses on the solution, not the problem, and provides practical and short-term well-being, has been started to be used in the management of violent behavior and anger.

SFA is an initiative that respects individuals and believes in their own resources and potential. In SFA, the problems of the individual are not examined, the resources and strengths of the individual are determined. Access to these resources provides an important opportunity for the individual to discover their skills and abilities. SFA meets the values and principles of mental health and psychiatric nursing on a common ground, as the individual searches for the skills and power resources that the individual will use in the process of change. Psychiatric nurses focus on good and working solutions and on the moments when the problem will not happen, instead of focusing on the problem and deficiencies, in order to contribute to the individual's adaptation and solution-generating skills. With this support, the individual is provided with an important opportunity to realize their personal characteristics and develop their social skills. Although SFA can be applied to all age groups, the most effective evidence-based studies are those in which children and adolescents participate.

In this study, unlike other studies, it is aimed to contribute to the literature by examining the effect of SFA on improving anger management and reducing the level of violence in adolescents. SFA intervention can be used as a nursing intervention in adolescents with low anger control and high tendency to violence. When psychiatric nurses use SFA principles and practices; It contributes in areas such as protecting and improving adolescent health, reducing violence and aggression behaviors, providing anger management, strengthening talents, skills and capacities, and improving in case of illness, in order to create healthier generations free from violence.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* High tendency to violence score
* High trait anger score
* Anger control score is low

Exclusion Criteria:

* With a psychiatric diagnosis
* Diagnosed with an organic chronic disease
* Participating in any support group or psychotherapy
* Students with special educational needs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Trait Anger and Anger Expression level in adolescents | 4 weeks after solution-focused intervention
  The primary outcome of this study was the mean adolescents trait anger level and Anger Expression level of the at 1 week and 4 weeks after solution-focused intervention. These levels of adolescents were evaluated using the State-Trait Anger Expression Scale (STAXI). The scale comprises 34 items and 2 sub-dimensions. The first 10 items of the scale indicate trait anger. The highest score that can be obtained from the Trait Anger scale is 40 and the lowest score is 10. A high score indicates that the individual has a high level of trait anger.
  The 24 items after the first 10 items consist of items measuring anger expression styles. 8 of these items are related to keeping anger in, 8 of them are related to keeping anger out, and the remaining 8 are related to anger control. The lowest score that can be obtained from each of these 3 sub-dimensions is 8, and the highest score is 32. A high score indicates high anger-in and anger-out levels, while low anger control.
Violent Behavior level in adolescents | 4 weeks after solution-focused intervention
  The other main outcome of the study was the adolescents' violence tendency level at 1 week and 4 weeks after the solution-focused intervention. The violence tendency level of the adolescents was evaluated using the Violence Tendency Scale (VTS). The scale consists of 20 items. The lowest score that can be obtained from the scale is 20, and the highest score is 60. A high score indicates that the level of violence tendency of the individual is also high.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Akbaş, RN, PhD, Principal Investigator — Pamukkale University; Gülay Taşdemir Yiğitoğlu, RN, PhD, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Kınıklı Campus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No